CLINICAL TRIAL: NCT05910957
Title: Multi-Omic, Clinomic and Digitomic Attributes of Major Depression for Integrative Analytics: the MACADAMIA Pilot Study
Brief Title: Multi-Omic, Clinomic and Digitomic Attributes of Major Depression for Integrative Analytics
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Florida State University (Other)
Responsible Party: Principal Investigator, Mohit Chauhan, M.B.B.S., Principal Investigator, Mayo Clinic
Other Study IDs: 23-002931
Record Dates: First submitted 2023-06-11; First posted 2023-06-20 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder; Unipolar, Non-psychotic Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study will collect 20 mL of blood for biomarker discovery efforts. Specifically, this study will collect and store blood samples that will be used in the future to derive C-reactive protein (CRP) levels, genome-wide genomics, proteomics, metabolomics, and exposomics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-depressed controls: Subjects without depression will fill out questionnaires about their general health and wellbeing, quality of life, mental health, emotional health, suicide risk, support system, and childhood experiences. Smartwatch data will also be collected to monitor step count, sleep quality, heart rate (resting and active), and activity rates.
- Antidepressant-treated adults: Subjects diagnosed with depression will fill out questionnaires about their general health and wellbeing, quality of life, mental health, emotional health, suicide risk, support system, and childhood experiences. Smartwatch data will also be collected to monitor step count, sleep quality, heart rate (resting and active), and activity rates.

SUMMARY:
The purpose of this research is to see if information from blood and data from smartwatches can be combined to help diagnose depression and determine if transitions between active depression and treated depression can be predicted.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the BROWNIE study.
* DSM-5 diagnostic criteria are met for unipolar, non-psychotic MDD (excluding controls).
* A score of > 10 on the QIDS-C and QIDS-SR (equivalent to 13 or greater on HAM-D17) given that when medication exceeds the effect of placebo in primary care participants have a HAM-D17 >12 (excluding controls).
* Antidepressant treatment is deemed appropriate by a study clinician (excluding controls).
* Smart watch wear time is at least 70% during their participation in the BROWNIE study.

Exclusion Criteria:

* Subjects with medical contraindications that preclude treatment with study drugs will be excluded.
* Patients with schizophrenia, schizoaffective disorder, or who have bipolar I or II disorder (or another specified or unspecified bipolar spectrum disorder) will be excluded because they have a primary psychiatric condition that requires a different initial treatment.
* Subjects currently on antidepressant medication with subtherapeutic results in terms of depression management will undergo a medication taper and discontinuation prior to initiation of a new study medication. The subject will be closely monitored by the study clinician during the medication taper and discontinuation phase. The medication taper is left up to the study clinician's discretion. Study subjects who cannot be safely tapered from their medication or experience adverse effects during the taper will be excluded from the study.
* Subjects who have an active substance use disorder will be excluded. An active substance use disorder will be defined as meeting DSM-5 diagnostic criteria for any active substance use disorder. Persons meeting DSM-5 diagnostic criteria for a substance use disorder in full remission (>12 months) and a negative urine drug of abuse screen at the screening visit or before the baseline study visit will be considered eligible. Persons with a positive urine drug of abuse screen may participate in the study if they do not meet DSM-5 diagnostic criteria for a substance use disorder.
* Subjects unable to give informed consent or who are unwilling or unable to comply with study requirements are excluded.
* Pregnant subjects will be excluded.
* Subjects who are currently breastfeeding and who plan to continue breastfeeding will be excluded.
* Subjects who are psychiatrically hospitalized or in a mental health crisis requiring urgent care or psychiatric hospitalization.
* Study subjects currently on antipsychotic medications (e.g., typical, and atypical antipsychotic drugs) taken for primary psychotic illness or affective psychosis will be excluded.
* Study subjects taking mood stabilizing agents (e.g., lithium, carbamazepine, valproate, lamotrigine, gabapentin, or other anticonvulsants) taken specifically for bipolar spectrum disorders are not eligible for participation.

Ages: 20 Years to 62 Years | Sex: All
Age Groups: Adult
Study Population: Subjects will be recruited from an ongoing cohort study at Mayo Florida "Wearable Augmented Prediction of Burnout in Nurses: A Synergy of Engineering, Bioethics, Nursing and Wellness Sciences" (BROWNIE Study)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2026-06-06 (Estimated); Study Completion 2026-12-06 (Estimated)

PRIMARY OUTCOMES:
Change in Quick Inventory of Depressive Symptoms-Clinician Rated (QIDS-CR) scale | Baseline, 4 weeks, and 8 weeks
  The Quick Inventory of Depressive Symptoms-Clinician Rated is used for rating the severity of depressive symptoms. Possible scores range from 0 to 27, with higher scores indicating greater severity of depression.

SECONDARY OUTCOMES:
Change in Hamilton Depression Rating Scale | Baseline, 4 weeks, and 8 weeks
  The Hamilton Depression Rating Scale is used for rating the severity of depressive symptoms. Possible scores range from 0 to 50, with higher scores indicating greater severity of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Chauhan, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No